CLINICAL TRIAL: NCT06079086
Title: Evaluation of the Clinical Evolution of Breast Increase Using Prostheses With Textured Silicone Envelope and Prostheses With Silicone Velvet Envelope
Brief Title: Evaluation of the Clinical Evolution of Breast Increase Using Prostheses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lifesil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LIFESIL_001
Record Dates: First submitted 2023-10-03; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Breast Augmentation; Mammoplasty

STUDY DESIGN:
Intervention Model Description: velvet/silicone foam envelope silicone with textured envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - group with textured envelope (Active Comparator): Group A - group with textured envelope
  Interventions: Device: Breast Implants Lifesil
- Group B - group with velvet/silicone foam envelope (Active Comparator): Group B - group with velvet/silicone foam envelope
  Interventions: Device: Breast Implants Lifesil

INTERVENTIONS:
Device: Breast Implants Lifesil — The surgery is performed through an incision (4 cm) in the inframammary fold and displacement in the supra-muscular plane, creation of a pocket for the inclusion of the prosthesis, followed by strict hemostasis and washing with an antibiotic solution. Placement of the prosthesis by digital maneuver and closure in layers using absorbable synthetic 4-0 polycaprolactone suture. Afterwards, an occlusive dressing is applied to the surgical wound. IV antibiotics (cephalosporin) 1g are administered at the beginning of surgery, followed by repeat/booster doses every 6 hours in the first 24 hours. Analgesic and anti-inflammatory medications are administered, varying according to each patient's restrictions.

SUMMARY:
The breasts are paired, superficial organs with relative symmetry. They particularly characterize femininity as an erogenous area, in addition to playing an extremely important role in a woman's body aesthetics. Breast augmentation surgery aims to add volume or restore breast volume lost post-pregnancy or weight loss, often establishing a balance in the body silhouette and increasing self-esteem. Breast implants cause an inflammatory reaction with the consequent formation of a fibrous capsule around the implant, which can evolve with different degrees of contraction.

Different factors are involved with the formation and intensity of the peri-prosthetic capsule: presence of hematoma, sub-clinical infection, silicone leakage, type of prosthetic envelope, plane/site of prosthesis placement, immune response, among others. The involvement of the envelope texture proved to be a major factor in reducing the formation of capsular contracture, which was clearly evident when covering with polyurethane foam was used. It is estimated that this reduction is due to the three-dimensional structure obtained with this configuration, which would result in a smaller vector resultant of contraction of the capsular fibers.

Aiming to obtain less capsular contracture, a silicone prosthesis with a velvet/silicone foam envelope was developed, which theoretically would have the advantage of the velvet/foam structure similar to polyurethane without, however, presenting negative aspects such as degradation, inflammation and eventual toxicity of catabolites. In this way, it is expected to prove the best postoperative evolution regarding the use of silicone prostheses with velvet/silicone foam coverage, highlighting the maintenance of the breast position over time. Furthermore, to intend to verify whether the velvet/silicone foam coverage determines a lower incidence of capsular contracture compared to the textured envelope. To this end, evaluation will be carried out through clinical examination and evaluation of digital photographic images taken pre-operatively, 30, 120, and 360 days post-operatively.

After a long postoperative period (approximately 9 years), a late follow-up will be carried out with the patients with clinical evaluation and a satisfaction questionnaire.

DETAILED DESCRIPTION:
The breasts are paired, superficial organs with relative symmetry. They particularly characterize femininity as an erogenous area, in addition to playing an extremely important role in a woman's body aesthetics. Breast augmentation surgery aims to add volume or restore breast volume lost post-pregnancy or weight loss, often establishing a balance in the body silhouette and increasing self-esteem. Breast implants cause an inflammatory reaction with the consequent formation of a fibrous capsule around the implant, which can evolve with different degrees of contraction.

Different factors are involved with the formation and intensity of the peri-prosthetic capsule: presence of hematoma, sub-clinical infection, silicone leakage, type of prosthetic envelope, plane/site of prosthesis placement, immune response, among others. The involvement of the envelope texture proved to be a major factor in reducing the formation of capsular contracture, which was clearly evident when covering with polyurethane foam was used. It is estimated that this reduction is due to the three-dimensional structure obtained with this configuration, which would result in a smaller vector resultant of contraction of the capsular fibers.

Aiming to obtain less capsular contracture, a silicone prosthesis with a velvet/silicone foam envelope was developed, which theoretically would have the advantage of the velvet/foam structure similar to polyurethane without, however, presenting negative aspects such as degradation, inflammation and eventual toxicity of catabolites. In this way, it is expected to prove the best postoperative evolution regarding the use of silicone prostheses with velvet/silicone foam coverage, highlighting the maintenance of the breast position over time. Furthermore, to intend to verify whether the velvet/silicone foam coverage determines a lower incidence of capsular contracture compared to the textured envelope. To this end, evaluation will be carried out through clinical examination and evaluation of digital photographic images taken pre-operatively, 30, 120 and 360 days post-operatively.

After a long postoperative period (approximately 9 years), a late follow-up will be carried out with the patients with clinical evaluation and a satisfaction questionnaire.

It is expected to demonstrate better postoperative evolution when using silicone prostheses with velvet/silicone foam coverage, highlighting the maintenance of position and less capsular contracture. To evaluate the participants' satisfaction with the silicone prosthesis after a prolonged post-operative period, through a satisfaction questionnaire, where the questions will be applied in a face-to-face consultation with the study doctor, who will also evaluate the participants' clinical conditions. Data will be obtained to evaluate the safety and efficacy of the implant over the long term of implantation.

ELIGIBILITY:
Inclusion Criteria:

* who present complaints of hypomastia of different etiologies (constitutional hypotrophy, post-weight loss, post-breastfeeding

Exclusion Criteria:

* who have already had a prosthesis included before the clinical study and/or for prosthesis exchange
* with sequelae of mastectomy with loss of architecture of the breast region and requiring additional surgeries (flaps, grafts)
* with decompensated chronic disease
* pregnant or postpartum women
* minors, vulnerable with mental problems
* patients who have breast ptosis and require mastopexy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 1 year
  Evaluate the possible occurrence of capsular contracture, maintenance of the position of the prosthesis and shape of the breasts postoperatively at 30, 120 and 360 days. Through clinical examination and standardized photographic documentation.

SECONDARY OUTCOMES:
Evaluate the long-term safety and effectiveness of prostheses (8-9 years) | 8-9 years
  To evaluate the safety and effectiveness of prostheses in the long term (8-9 years), through a questionnaire applied in a clinical consultation, with a late post-operative follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Kharmandayan, PhD, Principal Investigator — University of Campinas, Brazil

IPD SHARING:
Plan to Share IPD: No